CLINICAL TRIAL: NCT00341016
Title: Scientific Protocol for the Study of Leukemia and Other Hematologic Diseases Among Clean-up Workers in Ukraine Following the Chernobyl Accident
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999996030; OH96-C-N030; NCT00558974 (obsolete NCT alias); NCT01338233 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Leukemia
Keywords: Radiation
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort of Chernobyl cleanup workers (liquidators) in Ukraine: Cases with leukemia and related diseases, and matched controls in the cohort

SUMMARY:
Leukemia holds a special place in the study of radiation-related cancer because bone marrow is one of the tissues most sensitive to the carcinogenic effect of ionizing radiation, radiogenic leukemia has the shortest latent period among radiation-induced cancers, and its appearance suggests that solid tumors may follow. These same characteristics also contribute to its considerable significance in radiation protection. There are, nevertheless, important gaps in existing knowledge of radiation-induced leukemia, gaps that derive from characteristics of the study of the atomic bombing of Hiroshima and Nagasaki, and from studies of the effects of medical irradiation and studies of nuclear workers, these being the studies that have provided most of the information to date. These gaps include the presumed reduction in risk resulting from dose-fractionation and low dose-rate, and the time-response function in the first five years after exposure.

The primary objective of this study is to investigate leukemia risk as a function of such radiation; it would constitute the largest epidemiologic study conducted to date among working-age males, a group of particular concern in establishing occupational radiation safety standards. In addition, data on cases of multiple myeloma and myelodysplasia identified in the cohort will be collected to test the hypothesis of a dose related association between radiation and increased risk for each of these diseases.

The primary scientific objectives of the proposed study are to test the following hypotheses: (a) that there is a dose-related increase in risk of leukemia among these liquidators; (b) that the magnitude of any observed risk per unit dose is less than that seen in the atomic bomb survivors, exposed to essentially instantaneous radiation.

Subsidiary objectives include: (a) to investigate the nature of the dose-response relationship among liquidators and to identify modifiers of risk, including time since exposure, age at exposure, etc.; (b) to test the hypothesis that there is a dose-related increased risk of multiple myeloma; (c) to test the hypothesis that there is a dose-related increased risk of myelodysplasial; (d) to collect and store buccal cells from about 2,000 liquidators with a wide range of dose estimates extending to well over 1 Gy for possible use in future molecular studies of their DNA.

DETAILED DESCRIPTION:
Leukemia holds a special place in the study of radiation-related cancer because bone marrow is one of the tissues most sensitive to the carcinogenic effect of ionizing radiation. Radiogenic leukemia has the shortest latent period among radiation-induced cancers, and its appearance suggests that solid tumors may follow. These same characteristics also contribute to its considerable significance in radiation protection. There are, nevertheless, important gaps in existing knowledge of radiation-induced leukemia, gaps that derive from characteristics of the study of the atomic bombing of Hiroshima and Nagasaki, and from studies of the effects of medical irradiation and studies of nuclear workers; these are the studies that have provided most of the information to date. The gaps include the presumed reduction in risk resulting from dose-fractionation and low dose-rate, as well as the time- response function in the first five years after exposure. The study described herein is intended to fill those gaps.

The Chornobyl accident exposed hundreds of thousands of people to radiation, notably those involved in its cleanup operations. The second phase of a case-control study of ionizing radiation and leukemia is being conducted in a cohort of approximately 100,000 Ukrainian "liquidators" involved in cleanup work following the accident at the Chornobyl Nuclear Power Plant in northern Ukraine which occurred on April 26, 1986. The cohort is restricted to liquidators who first worked around the power plant between 1986 and 1990 and were residents, when first registered in the Chornobyl State Registry, in Kyiv City or in one of five oblasts (major civil divisions) that comprise the study area. This cohort, consisting of males of working age, received mean bone marrow doses of approximately 80-100 milli-gray (mGy) at low to moderate dose rates, with those sent earlier receiving the highest doses. The primary objective of this study is to investigate leukemia risk as a function of such radiation; it constitutes probably the largest epidemiologic study conducted to date among working-age males, a group of particular concern in establishing occupational radiation safety standards.

The primary scientific objectives of the proposed study are to evaluate whether there is a doserelated increase in risk of leukemia among these liquidators, and how it compares with the observed risk per unit dose seen in the atomic bomb survivors, exposed to essentially instantaneous radiation. A secondary objective is to identify any modifiers of risk, including time since exposure, age at exposure, etc.

The field work for the second phase of the study, with an extended case ascertainment for 2001 through 2006 has been complated. As a result of the second phase, a total of75 confirmed cases of leukemia and 12 cases of multiple myeloma have been ascertained. We are currently in the process of database construction, dosimetric calculation for data analyses for leukemia, and manuscript preparation.

The small sub-study on uncertainties associated with human factors is to be started upon SSIRB approval.

ELIGIBILITY:
* INCLUSION CRITERIA:

We intend to include in the proposed study all 350 clean-up workers with "historical" records and 150 proxies to be identified by the liquidators; however, we anticipate a considerable number of them will not be available for the study due to deaths, not being able to be traced, no response, refusals, etc. The study subjects will be interviewed in person. All study subjects are males, median age of early liquidators is 64 y while for clean-up workers sent to mission is about 61 years.

EXCLUSION CRITERIA:

Excluded from the study will be those who have been found to be deceased, cannot be located, refuse to participate in the study, or do not provide informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ukrainian Chernobyl cleanup workers ("liquidators") approx. 100,000 persons
Sampling Method: Probability Sample
Enrollment: 1779 (Actual)
Dates: Start 1996-08-26 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to investigate leukemia risk as a function of radiation ionizing radiation from occupational exposure (Chernobyl nuclear power plant) | time of interview
  Estimated risk of leukemia related to radiation exposure

CONTACTS AND LOCATIONS:
Overall Officials: Kiyohiko Mabuchi, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Research Center for Radiation Medicine, Kiev, Ukraine

REFERENCES:
- [Background] Gudzenko N, Hatch M, Bazyka D, Dyagil I, Reiss RF, Brenner A, Chumak V, Babkina N, Zablotska LB, Mabuchi K. Non-radiation risk factors for leukemia: A case-control study among chornobyl cleanup workers in Ukraine. Environ Res. 2015 Oct;142:72-6. doi: 10.1016/j.envres.2015.06.019. Epub 2015 Jun 24. PMID 26117815
- [Background] Chumak VV, Romanenko AY, Voilleque PG, Bakhanova EV, Gudzenko N, Hatch M, Zablotska LB, Golovanov IA, Luckyanov NK, Sholom SV, Kryuchkov VP, Bouville A. The Ukrainian-American study of leukemia and related disorders among Chornobyl cleanup workers from Ukraine: II. Estimation of bone marrow doses. Radiat Res. 2008 Dec;170(6):698-710. doi: 10.1667/RR1403.1. PMID 19138037
- [Background] Zablotska LB, Bazyka D, Lubin JH, Gudzenko N, Little MP, Hatch M, Finch S, Dyagil I, Reiss RF, Chumak VV, Bouville A, Drozdovitch V, Kryuchkov VP, Golovanov I, Bakhanova E, Babkina N, Lubarets T, Bebeshko V, Romanenko A, Mabuchi K. Radiation and the risk of chronic lymphocytic and other leukemias among chornobyl cleanup workers. Environ Health Perspect. 2013 Jan;121(1):59-65. doi: 10.1289/ehp.1204996. Epub 2012 Nov 8. PMID 23149165